CLINICAL TRIAL: NCT04118842
Title: An Open-label, 3-period Fixed-sequence Study in Healthy Subjects to Assess the Pharmacokinetics of Savolitinib When Administered Alone and in Combination With Rifampicin
Brief Title: A Study in Healthy Subjects to Assess the Pharmacokinetics of Savolitinib When Administered Alone and in Combination With Rifampicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: D5084C00003
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumors
Keywords: Solid tumors; Small-molecule kinase inhibitor
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Savolitinib and/or Rifampicin (Experimental): Treatment Period 1 consists of 16 days starting with admission on Study Day -1, followed by a single dose administration of savolitinib on Day 1, followed by a washout period of at least 14 days. Subjects will be discharged from the Study Centre on Study Day 3, after the last PK sample is collected Treatment Period 2 consists of 6 days, starting with admission on Study Day 14, followed by QD dose administrations of rifampicin for 5 consecutive days (Study Day 15 to Study Day 19) Treatment Period 3 consists of 4 days, starting immediately after Treatment Period 2, comprising of a single dose administration of savolitinib on Study Day 20 and QD dose administration of rifampicin on Study Day 20 and Study Day 21. Subjects will be discharged from the Study Centre on Study Day 22, after the last PK sample is collected
  Interventions: Drug: Savolitinib; Drug: Rifampicin

INTERVENTIONS:
Drug: Savolitinib — Patients will receive a single dose on Study Day 1 and Study Day 20. Savolitinib will be administrated after a high fat, high calorie breakfast to reduce the risk of adverse events.
Drug: Rifampicin — Patients will receive Rifampicin once daily on Study Day 15, 16, 17, 18, 19, 20 and 21. Rifampicin will be administered 1 hour before breakfast.
  Other Names: Rifampin

SUMMARY:
This is a phase I, open-label, 3 treatment period, fixed-sequence study in healthy non-Japanese male subjects, aged 18 to 65 years (inclusive), performed at a single study centre. Treatment Period 1 will establish the single dose pharmacokinetic (PK) profile of savolitinib. Dosing of daily rifampicin during Treatment Period 2 will result in maximal induction of the CYP450 enzymes including CYP3A4. Treatment Period 3 will then establish the single dose PK profile of savolitinib under maximum CYP450 induction conditions. Comparison of the PK profile of savolitinib between Treatment Period 1 and Treatment Period 3 will quantify the effect of CYP450 enzyme induction.

DETAILED DESCRIPTION:
The treatment starts with a single dose of savolitinib (Treatment Period 1), followed by a washout period at least of 14 days after savolitinib dosing and before the start of Treatment Period 2, followed by rifampicin administration for 5 days (Treatment Period 2), and lastly, a combination of savolitinib + rifampicin (Treatment Period 3). Overall, all subjects will receive 2 single doses of 600 mg savolitinib and 7 daily doses of 600 mg rifampicin. Subjects will be resident in the study centre when receiving study drug administrations (savolitinib [Treatment Period 1], rifampicin [Treatment Period 2] and savolitinib+rifampicin [Treatment Period 3]). Subjects are required to fast overnight before each dosing day. Rifampicin will be administered 1 hour before breakfast with 240 mL water. The subjects will need to complete high-fat, high calorie breakfast before administration of savolitinib in Treatment Period 1, Day 1 (Study Day 1) and Treatment Period 3 Day 1 (Study Day 20).

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects should fulfil the following criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects with suitable veins for cannulation or repeated venipuncture: non Japanese male subjects aged 18 to 65 years (inclusive).
3. Have a body mass index between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
4. Alanine aminotransferase, AST and total bilirubin less than or equal to the upper limit of normal for the institution.
5. Have a calculated creatinine clearance greater than 80 mL/min using the Cockcroft-Gault formula at screening.
6. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this clinical study protocol.

Exclusion Criteria:

Subjects will not enter the study if any of the following exclusion criteria are fulfilled:

1. Healthy subjects of Japanese ethnicity and any healthy subject that has 1 parent or grandparent (maternal or paternal) of Japanese ethnicity.
2. History of any clinically significant disease or disorder which, in the opinion of the Principal Investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
3. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
5. Planned in-patient surgery, dental procedure or hospitalization during the study.
6. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the PI.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.
8. Abnormal vital signs, after 5 minutes supine rest, defined as any of the following:

(1) Systolic BP < 90 mmHg or ≥ 140 mmHg (2) Diastolic BP < 50 mmHg or ≥ 90 mmHg (3) Heart rate < 45 or > 85 beats per minute. 9 Any clinically important abnormalities in rhythm, conduction or morphology of the 12 lead resting ECG that may interfere with the interpretation of QTc interval changes. These include healthy subjects with any of the following:

1. Abnormal ST-T-wave morphology, particularly in the protocol defined primary lead (V2) or left ventricular hypertrophy.
2. PR interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
3. PR interval prolongation (> 200 ms). Intermittent second (Type 1 second degree block [Wenckebach Phenomenon] while asleep is not exclusive]) or third degree atrioventricular (AV) block, or AV dissociation.
4. Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre-excitation.
5. Mean resting correct QT interval (QTcF) > 450 ms for men on screening obtained from 3 ECGs or history or factors that may increase the risk of QTcF prolongation such as chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes (TdP).

10 Known or suspected history of drug abuse, as judged by the PI. 11 Current smokers or those who have smoked or used nicotine products within the previous 30 days.

12 History of alcohol abuse or excessive intake of alcohol as judged by the PI. 13 Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate,) as judged by the PI.

14 Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of the IMP.

15 Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first admission on Day -1.

16 Use of any prescribed or non-prescribed medication including antacids, analgesics (other than use of ibuprofen up to 72 hours before dosing day), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the first administration of the IMP or longer (5 times the half-life) if the medication has a long half-life. No medications known to prolong the QT/QTc interval and cause TdP are allowed.

17 Positive screen for drugs of abuse, cotinine (nicotine) and/or alcohol at screening and at admission to the Study Centre (Day -1 [Period 1] and Day 14 [Period 2]) to the Study Centre.

18 History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI.

19 History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to savolitinib or rifampicin.

20 Plasma donation within 1 month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.

21 Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.

Note: subjects consented and screened, but not enrolled in this study or a previous phase I study, are not excluded.

22 Involvement of any AstraZeneca, Parexel or study site employee or their close relatives 23 Subjects who have previously received savolitinib. 24 Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

25 Subjects who are vegans, vegetarians or have medical dietary restrictions and who are lactose intolerant.

26 Subjects who cannot communicate reliably with the PI. 27 Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

28 Subjects who wear soft contact lenses, unless the subject is prepared to refrain from wearing soft lenses throughout Period 2 until after the last PK sample collection in Period 3.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 40 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Savolitinib: Maximum plasma concentration (Cmax) ratios of geometric means of test treatment (savolitinib+rifampicin), relative to reference treatment (savolitinib alone) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To assess the effect of rifampicin on the PK of savolitinib
Area under the curve (AUC) ratios of geometric means of test treatment (savolitnib+rifampicin) relative to reference treatment (savolitinib alone) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To assess the effect of rifampicin on the PK of savolitinib

SECONDARY OUTCOMES:
Number of subjects with adverse events | Only SAEs at Screening; AEs from Study Days 1 to 34
  To assess the adverse events as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in systolic blood pressure (BP) | At Screening, and from Study Days 1 to 14 and Study Days 20 to 22
  To assess vital sign as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in diastolic BP | At Screening, and from Study Days 1 to 14 and Days 20 to 22
  To assess vital sign as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in pulse rate | At Screening, and from Study Days 1 to 14 and Study Days 20 to 22
  To assess vital sign as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in electrocardiograms (ECGs) (12-lead ECGs) | At Screening, and from Study Days 1 to 34
  To assess any clinically important abnormalities in cardiovascular function based on the 12-lead ECGs as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in physical examinations | At Screening, from Study Days -1 to 22 (brief) and Study Day 34
  To assess any clinically important abnormal findings in physical conditions as a variable of safety and tolerability of savolitinib in combination with rifampicin. The complete physical examinations will include an assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head and neck, lymph nodes, thyroid, musculoskeletal and neurological systems. The brief physical examinations will include an assessment of the general appearance, skin, abdomen, cardiovascular system and respiratory.
Number of subjects with abnormal findings in white blood cell (WBC) count | From Screening to Study Day 34
  To assess the WBC count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in red blood cell (RBC) count | From Screening to Study Day 34
  To assess the RBC count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in hemoglobin (Hb) | From Screening to Study Day 34
  To assess Hb as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in hematocrit (HCT) | From Screening to Study Day 34
  To assess HCT as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in mean corpuscular volume (MCV) | From Screening to Study Day 34
  To assess MCV as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in mean corpuscular hemoglobin (MCH) | From Screening to Study Day 34
  To assess MCH as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in mean corpuscular hemoglobin concentration (MCHC) | From Screening to Study Day 34
  To assess MCHC as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in neutrophils absolute count | From Screening to Study Day 34
  To assess the neutrophils absolute count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in lymphocytes absolute count | From Screening to Study Day 34
  To assess the lymphocytes absolute count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in monocytes absolute count | From Screening to Study Day 34
  To assess the monocytes absolute count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in eosinophils absolute count | From Screening to Study Day 34
  To assess the eosinophils absolute count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in basophils absolute count | From Screening to Study Day 34
  To assess the basophils absolute count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in platelets | From Screening to Study Day 34
  To assess platelets as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in reticulocytes absolute count | From Screening to Study Day 34
  To assess the reticulocytes absolute count as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in sodium | From Screening to Study Day 34
  To assess the clinical chemistry value (sodium) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in potassium | From Screening to Study Day 34
  To assess the clinical chemistry value (potassium) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in urea | From Screening to Study Day 34
  To assess the clinical chemistry value (urea) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in creatinine | From Screening to Study Day 34
  To assess the clinical chemistry value (creatinine) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in albumin | From Screening to Study Day 34
  To assess the clinical chemistry value (albumin) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in calcium | From Screening to Study Day 34
  To assess the clinical chemistry value (calcium) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in phosphate | From Screening to Study Day 34
  To assess the clinical chemistry value (phosphate) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in glucose (fasting) | From Screening to Study Day 34
  To assess the clinical chemistry value (glucose [fasting]) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in c-reactive protein (CRP) | From Screening to Study Day 34
  To assess the clinical chemistry value (CRP) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of participants with abnormal findings in liver enzymes | From Screening to Study Day 34
  To assess the clinical chemistry value of liver enzymes as a variable of safety and tolerability of savolitinib in combination with rifampicin. The laboratory variables to be measured are: alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), and gamma glutamyl transpeptidase (GGT)
Number of subjects with abnormal findings in total bilirubin | From Screening to Study Day 34
  To assess the clinical chemistry value (total bilirubin) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in unconjugated bilirubin | From Screening to Study Day 34
  To assess the clinical chemistry value (unconjugated bilirubin) as a variable of safety and tolerability of savolitinib in combination with rifampicin
Number of subjects with abnormal findings in urinalysis | From Screening to Study Day 34
  To assess the urinalysis as a variable of safety and tolerability of savolitinib in combination with rifampicin. The laboratory variables to be measured are protein, glucose, and blood.
Number of subjects with abnormal findings in urinalysis (microscopy) | From Screening to Study Day 34
  To assess the urinalysis microscopy (if positive for protein or blood) as a variable of safety and tolerability of savolitinib in combination with rifampicin. The laboratory variables to be measures are RBC, WBC, casts (cellular, granular, hyaline).
Savolitinib: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC[0-t]) ratios of geometric means of test treatment (savolitinib+rifampicin), relative to reference treatment (savolitinib alone) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To assess the effect of rifampicin on the PK of metabolites N-desmethyl savolitinib or 3-[(1S)-1-imidazo[1,2-a]pyridin-6-ylethyl]-5-(1H-pyrazol-4-yl)triazolo[4,5-b]pyrazine (M2) and 1-[(1S)-1-imidazo[1,2-a]pyridin-6-ylethyl]-6-(1 methylpyrazol-4-yl)triazolo[4,5-b]pyrazin-5-ol (M3)
M2 and M3: Cmax ratios of geometric means of test treatment (savolitinib+rifampicin), relative to reference treatment (savolitinib alone) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
M2 and M3: AUC ratios of geometric means of test treatment (savolitinib+rifampicin), relative to reference treatment (savolitinib alone) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
M2 and M3: AUC(0-t) ratios of geometric means of test treatment (savolitinib+rifampicin), relative to reference treatment (savolitinib alone) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: summary PK profiles and descriptive statistics of Cmax | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: summary PK profiles and descriptive statistics of AUC | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: summary PK profiles and descriptive statistics of AUC(0 t) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: Ratio of metabolite AUC to parent AUC (MRCAUC) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: Ratio of metabolite AUC(0-t) to parent AUC(0-t) (MRCAUC[0-t]) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: metabolite-to-parent ratios for Time to reach maximum observed plasma concentration (tmax) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: metabolite-to-parent ratios for Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2,λz) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: metabolite-to-parent ratios for terminal elimination rate constant (λz) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib: Apparent total body clearance of drug from plasms after extravascular administration (parent drug only)CL/F | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, when it is administered alone and in combination with rifampicin
Savolitinib, M2 and M3: Ratio of metabolite Cmax to parent Cmax (MRCmax) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib, M2 and M3 when savolitinib is administered alone and in combination with rifampicin
Savolitinib: Apparent volume of distribution during the terminal phase after extravascular administration (parent drug only) (Vz/F) | Treatment Period 1 (Study Days 1 to 14) and Treatment Period 3 (Study Days 20 to 22) at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after study drug administration
  To describe the PK parameters and the PK profiles for savolitinib it is administered alone and in combination with rifampicin

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States